CLINICAL TRIAL: NCT00770055
Title: Internet Use Among Women With Recurrent Breast Cancer
Brief Title: Internet Use Among Women With Recurrent Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Deborah Toppmeyer, MD, Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School
Organization: Rutgers, The State University of New Jersey (Other)
Purpose: Health Services Research
Other Study IDs: CDR0000592835; P30CA072720 (NIH); CINJ-000102; CINJ-IRB-3879
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Other: survey administration
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Gathering information about patients with breast cancer over time may help doctors learn more about a patient's use of the internet to find information about treatment, symptom management, and emotional support.

PURPOSE: This clinical trial is studying internet use among women with recurrent metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To document the proportion of women who use the internet to access treatment and symptom management information and to seek emotional support after diagnosis of metastatic recurrent breast cancer.
* To evaluate the association of treatment stage and effectiveness with internet use.
* To evaluate the association of individual differences in patients' demographics, beliefs, emotional functioning, and social and professional support with internet use.
* To evaluate the association of patients' use of the internet to seek resources with their beliefs, emotional functioning, and relationship functioning.

OUTLINE: Patients undergo assessments consisting of paper and pencil questionnaires at four time points. The timing of these assessments is linked to the patient's treatment course and her presumed need to access internet resources for information on cancer, treatment, symptom management, and emotional support. Patients who discontinue regular care at the Cancer Institute of New Jersey site during the course of the study may complete study assessments through phone interviews conducted by a member of the study team.

Patients undergo a baseline survey prior to deciding on a treatment course for their newly progressive disease. Patients complete the first part of the survey to provide information on demographics, beliefs about cancer, mood states, somatic symptoms, and available resources for cancer information and emotional support. Patients complete the second part of the survey, if they have used the internet previously to obtain information and resources about cancer or if they have received cancer information that someone else located on the internet for them, which inquires about patients' internet use, any internet resources they have received from family members, friends, or other people they know, and their own evaluation of these internet resources. Patients undergo the second study assessment after completion of the first course of treatment and prior to initiating course 2 (i.e., 3 to 4 weeks after initiating treatment). The third study assessment occurs within the first 2 weeks after the medical oncologist's first evaluation of treatment response (i.e., 6-9 weeks after initiating treatment). The fourth assessment occurs after the medical oncologist's second evaluation of the patient's response to treatment, following tumor re-staging.

Patients complete several questionnaires during these assessments to provide information about personal characteristics (demographics, physical and psychological well-being, beliefs about cancer and treatment, optimism), social and healthcare networks (perceived social support, social network composition, beliefs about treatment team), and outcomes (use of non-internet cancer information, use of the internet for cancer resources, use of interactive technologies, communication with treatment team and family, evaluation of internet resources).

The following information is extracted from the patients' medical record: stage and node status at primary diagnosis, previous oncology surgeries, previous adjuvant treatments, current menopausal status, treatment at time of recurrence, disease free interval, site(s) of metastasis, and response to current treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of recurrent breast cancer meeting either of the following criteria:

  * Newly diagnosed metastatic disease
  * Recently diagnosed as progressive disease after stable metastatic disease for at least 6 months

    * Must have received the same treatment for metastatic breast cancer for at least 3 months

      * Have received no treatment for progressive disease OR have begun treatment for progressive disease within the past month
* Patient at the Cancer Institute of New Jersey in New Brunswick or Hamilton, New Jersey
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Able to speak and write English
* Free of diseases and cognitive impairments that would interfere with comprehension of the survey instruments or ability to provide informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2001-11; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Use of non-internet cancer information
Use of the internet for cancer resources
Use of interactive technologies
Communication with treatment team and family members
Evaluation of internet resources
Changes in internet use over the course of treatment
Cross-sectional associations between patients' internet use and their individual, social, and professional network characteristics
Internet use and changes in patients' beliefs and emotional functioning

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Toppmeyer, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States